CLINICAL TRIAL: NCT00001032
Title: A Phase II Study to Evaluate Pharmacokinetics, Safety, Tolerance and Activity of Dideoxycytidine (ddC) Administered in Combination With Zidovudine (AZT) in Stable, AZT-Treated Pediatric Patients With HIV Infection
Brief Title: A Study of Dideoxycytidine Plus Zidovudine (AZT) in HIV-Infected Children Who Have Taken AZT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 190; 11165 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
PRIMARY: To determine safety, tolerance, and pharmacokinetics of zidovudine (AZT) and zalcitabine (dideoxycytidine; ddC) when given in combination in clinically stable AZT-treated children.

SECONDARY: To compare combination therapy with mono drug therapy for antiviral activity and laboratory markers of disease progression, as determined by virologic and immunologic determinations. To evaluate the influence of combination therapy on disease progression as determined by evaluation of clinical criteria.

In children currently being treated with AZT, it is unknown whether the addition of another antiretroviral agent such as ddC would help increase efficacy and tolerance. This study will examine the possible advantages of combination AZT/ddC therapy over monotherapy with AZT alone.

DETAILED DESCRIPTION:
In children currently being treated with AZT, it is unknown whether the addition of another antiretroviral agent such as ddC would help increase efficacy and tolerance. This study will examine the possible advantages of combination AZT/ddC therapy over monotherapy with AZT alone.

Patients are stratified according to duration of ongoing AZT therapy and are randomized to receive AZT either alone or in combination with ddC. Patients receive therapy until the last patient enrolled completes 32 weeks of therapy. The study may be extended for two additional 32-week periods on an optional basis.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* Intravenous and/or intramuscular immunoglobulin.
* Acyclovir (no more than 30 mg/kg/day PO).
* Ketoconazole (no more than 10 mg/kg/day).
* Nystatin.
* Aspirin, acetaminophen, nonsteroidal anti-inflammatory drugs, sedatives, and barbiturates, not to exceed 72 hours.
* Isoniazid in combination with pyridoxine, provided there is no evidence of peripheral neuropathy.
* Trimethoprim / sulfamethoxazole.
* Amphotericin B (no more than 1 mg/kg for 5 days/week).
* Aerosolized ribavirin for bronchiolitis.
* Hematopoietic agents.
* Other drugs with little nephro-, hepato-, or cytotoxicity.
* Nutritional support for HIV wasting syndrome or malnutrition.

Patients must have:

* HIV infection.
* Ongoing stable AZT therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Disease progression while on AZT, to the extent that the patient meets the criteria for advanced disease protocols.
* Known allergy or sensitivity to ddC.
* Cardiomyopathy.

Concurrent Medication:

Excluded:

* Biologic modifiers other than IVIG, steroids, or hematopoietic agents.
* Investigational medications unless approved by protocol chair.
* Medications known to cause pancreatitis (unless ddC is interrupted while these medications are given).

Patients with the following prior conditions are excluded:

* History of intolerance or toxicity to AZT.
* History of symptomatic pancreatitis.
* History of peripheral neuropathy or abnormal nerve conduction velocity test.

Prior Medication:

Excluded:

* Antiretroviral agents other than AZT within 2 weeks of study entry.

Required:

* Ongoing stable AZT therapy for more than 6 weeks duration.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180
Dates: Study Completion 1995-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Pahwa, Study Chair; SS Bakshi, Study Chair
Locations (47):
- United States (44):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - San Francisco Gen. Hosp., San Francisco, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Connecticut Health Ctr., Dept. of Ped., Farmington, Connecticut
  - Yale Univ. School of Medicine - Dept. of Peds., Div. of Infectious Disease, New Haven, Connecticut
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Univ. of Maryland Med. Ctr., Div. of Ped. Immunology & Rheumatology, Baltimore, Maryland
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - Children's Hospital at Albany Medical Center, Dept. of Peds., Albany, New York
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Metropolitan Hosp. NICHD CRS, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds., Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Bakshi SS, Britto P, Capparelli E, Mofenson L, Fowler MG, Rasheed S, Schoenfeld D, Zimmer B, Frank Y, Yogev R, Jimenez E, Salgo M, Boone G, Pahwa SG. Evaluation of pharmacokinetics, safety, tolerance, and activity of combination of zalcitabine and zidovudine in stable, zidovudine-treated pediatric patients with human immunodeficiency virus infection. AIDS Clinical Trials Group Protocol 190 Team. J Infect Dis. 1997 May;175(5):1039-50. doi: 10.1086/520351. PMID 9129064
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891